CLINICAL TRIAL: NCT01298583
Title: Ankle Tracking Training in Stroke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0508M72871
Record Dates: First submitted 2011-02-16; First posted 2011-02-17 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ankle tracking (Experimental): subjects track a target with ankle movement
  Interventions: Behavioral: ankle tracking training
- ankle movement (No Intervention)

INTERVENTIONS:
Behavioral: ankle tracking training — one group will use the ankle for tracking, the other group will use the ankle for simple movement
  Arms: ankle tracking

SUMMARY:
The purpose of this study is to compare the improvement in ankle control and brain activation in subjects with stroke resulting from two different forms of telerehabilitation: tracking training, emphasizing accurate movements, versus movement training, involving simple movements.

Hypotheses:

1. The Track group will show greater improvement in ankle range of motion compared to the Move group.
2. The Track group will show greater improvement in ankle tracking accuracy and greater changes in fMRI (increase in relative volume of activation for ipsilesional sensorimotor cortex, increase in laterality index, and decrease in blood-oxygen-level-dependent (BOLD) signal intensity index) compared to Move group.
3. The Track group will show greater improvement in tracking accuracy at an untrained joint (knee) compared to the Move group.
4. The Track group will show greater improvement in standing balance.
5. The Track group will show greater improvement in walking speed and ankle dorsiflexion during gait compared to the Move group.

ELIGIBILITY:
Inclusion Criteria:

1. Single stroke with an ischemic infarct.
2. Between 18 and 85 years of age.
3. Time since stroke onset must be >6 months.
4. Cannot be receiving any rehabilitation therapy.
5. Impaired ankle dorsiflexion/plantarflexion but at least 10 degrees of active motion.
6. Cognition level must be at least 24 out of 30 on the Mini-Mental Examination 7. Able to ambulate at least 100 feet independently. training.

Exclusion Criteria:

1. Cannot have any neuromuscular disorder other than stroke that impairs ankle motion.
2. Cannot have an executive function score on Stroop Interference Test of <37.
3. Cannot have a score on the Beck Depression Inventory of >10.
4. Cannot have ataxia, apraxia, receptive aphasia, hemi-neglect, or severe visual field cut .
5. Cannot be pregnant nor have indwelling metal or medical devices incompatible with fMRI.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
ankle range of motion | Measurement at pretest, posttest and followup

CONTACTS AND LOCATIONS:
Overall Officials: James Carey, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Deng H, Durfee WK, Nuckley DJ, Rheude BS, Severson AE, Skluzacek KM, Spindler KK, Davey CS, Carey JR. Complex versus simple ankle movement training in stroke using telerehabilitation: a randomized controlled trial. Phys Ther. 2012 Feb;92(2):197-209. doi: 10.2522/ptj.20110018. Epub 2011 Nov 17. PMID 22095209